CLINICAL TRIAL: NCT00195455
Title: A Prospective Open Label Study to Evaluate Vasomotor Symptoms Control and Bleeding Patterns With a Continuous Regimen of a New Progestin Trimegestone 0.125 mg and 17 b Estradiol 1 mg (Totelle),as HT on Postmenopausal Women
Brief Title: Study Evaluating Estradiol/Trimegestone in Vasomotor Symptoms (VMS) in Post-Menopausal Women.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0753T-101538
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2007-12-20 (Estimated); Status verified 2007-12

CONDITIONS: Postmenopause
Keywords: Postmenopause
MeSH Terms: interventions — trimegestone

INTERVENTIONS:
Drug: Trimegestone
Drug: 17b Estradiol

SUMMARY:
The purpose of this study is to evaluate vasomotor symptoms (VMS) control of the continuous regimen 17 b estradiol/trimegestone combination.

ELIGIBILITY:
Inclusion Criteria:

* Generally healthy postmenopausal women 45 to 55 years of age inclusive, with at least 1 year of natural occurring amenorrhea, with vasomotor symptoms, with at least 4 hot flushes per day
* Intact uterus

Exclusion Criteria:

* Known or suspected breast carcinoma or estrogen-dependent neoplasm
* Undiagnosed abnormal genital bleeding

Ages: 45 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 133 (Estimated)
Dates: Start 2005-02; Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
To assess vasomotor symptoms control with a continuous regimen of 17 b estradiol 1mg and Trimegestone (TMG) 0.125 mg.

SECONDARY OUTCOMES:
Study bleeding patterns throughout the treatment period (6 months)
Evaluate changes in the Menopause-Specific Quality of Life Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer; Trial Manager, Principal Investigator — For Mexico, gomezlj@wyeth.com
Locations (3):
- Mexico (3):
  - Guadalajara, Jalisco
  - Monterrey, N.L.
  - Mexico City